CLINICAL TRIAL: NCT03969953
Title: Treatment of Cardiovascular Disease With Low Dose Rivaroxaban in Advanced Chronic Kidney Disease
Acronym: TRACK
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Emerald Clinical Inc. (Industry); Bayer (Industry); Central Hospital, Nancy, France (Other); King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0040139
Record Dates: First submitted 2019-05-27; First posted 2019-05-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Diseases; Dialysis-dependent Kidney Failure; Cardiovascular Disease
Keywords: Rivaroxaban
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: The TRACK trial is an investigator-initiated, multicentre, prospective, randomised, quadruple-blind (participant, healthcare provider, data collector, outcomes assessor), placebo-controlled trial. The trial will test for the superiority of the trial intervention using a 1:1 allocation to parallel trial groups, on the basis of a pre-specified number of primary outcomes events.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple-blind, Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban 2.5mg, twice daily.
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet
- Placebo (Placebo Comparator): Matched placebo, twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — Rivaroxaban is an orally administered selective direct factor Xa inhibitor.
  Other Names: Xarelto
  Arms: Rivaroxaban
Other: Placebo — Rivaroxaban matched placebo
  Arms: Placebo

SUMMARY:
The TRACK trial is an investigator-initiated, multicentre, prospective, randomised, quadruple-blind (participant, healthcare provider, data collector, outcomes assessor), placebo-controlled trial. TRACK is a global trial and will be conducted in renal units that provide comprehensive CKD care. Approximately 2000 participants will be recruited.

The TRACK trial will assess a strategy of administering low dose rivaroxaban to reduce the risk of major adverse cardiac event (MACE) in people with Chronic Kidney Disease (CKD) stages 4 or 5 or dialysis-dependent kidney failure, and elevated cardiovascular (CV) risk (marked by a history of CAD or PAD, or non-haemorrhagic non-lacunar stroke OR diabetes mellitus OR age ≥65 years).

DETAILED DESCRIPTION:
Background and Rationale Chronic Kidney Disease (CKD) is a major international health burden. Despite the unacceptably high burden of cardiovascular disease (CVD) and associated mortality, trial-data on the management of CVD in people with advanced stages of CKD and dialysis-dependent kidney failure are sparse. Risk of bleeding in CKD and dialysis-dependent kidney failure is increased when compared to the general population. Anticoagulant agents, such as rivaroxaban, are a core intervention in the prevention of CVD in the general population. Nevertheless, to mitigate trial risks, 90% of the trials evaluating this form of intervention exclude these patient populations.

The TRACK trial will evaluate the effect of low dose rivaroxaban in patients with CKD dialysis-dependent kidney failure. Other trials have demonstrated that rivaroxaban reduces the risk of major cardio-vascular outcomes in high risk patients, and the limited data showed that CKD status did not significantly affect this result.

Hypothesis Compared to placebo, low dose rivaroxaban reduces the risk of major adverse cardiac event (MACE) in people with CKD stages 4 or 5 or dialysis-dependent kidney failure, and elevated cardiovascular (CV) risk (marked by a history of CAD or PAD, or non-haemorrhagic non-lacunar stroke OR diabetes mellitus OR age ≥65 years).

Objectives The primary objective is to determine whether low dose rivaroxaban, compared to placebo, significantly reduces the risk of a composite outcome of;

* CV death,
* non-fatal myocardial infarction,
* stroke, or
* peripheral artery disease (PAD) events

in people with CKD stages 4 or 5 or dialysis-dependent kidney failure, and an elevated CV risk (marked by a history of CAD or PAD, or non-haemorrhagic non-lacunar stroke OR diabetes mellitus OR age ≥65 years).

A full list of secondary objectives are detailed in the protocol, and include identifying risk reduction in the treatment group, and whether this treatment is cost effective.

Methodology The TRACK trial is an investigator-initiated, multicentre, prospective, randomised, quadruple-blind (participant, healthcare provider, data collector, outcomes assessor), placebo-controlled trial. The trial will test for the superiority of the trial intervention using a 1:1 allocation to parallel trial groups, on the basis of a pre-specified number of primary outcomes events.

This is a global trial and will be conducted in renal units that provide comprehensive CKD care. Approximately 2,000 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* People able to provide informed consent who meet all of the following inclusion criteria:

  1. Age ≥18 years,
  2. Kidney Failure on haemodialysis or peritoneal dialysis, or CKD stage 4 or 5 (eGFR ≤29 mL/min/1.73 m2) not receiving renal replacement therapy,
  3. Elevated cardiovascular risk, defined by at least one of the following:

     1. History of Coronary Artery Disease (CAD) or PAD or non-haemorrhagic non-lacunar stroke, or
     2. Diabetes mellitus, or
     3. Age ≥65 years.

Exclusion Criteria:

* Potential participants must have none of the following exclusion criteria at the time of study enrolment:

  1. Mechanical/prosthetic heart valve (does not include bioprosthetic valves that do not require therapeutic anticoagulation),
  2. Indication for, or contraindication to, anticoagulant therapy,
  3. High bleeding risk including any coagulopathy,
  4. Lesion or condition considered to be a significant risk of major bleeding,
  5. Major bleeding episode in the 30 days prior to study enrolment, or any active and clinically significant bleeding,
  6. Current treatment with P2Y12 inhibitors/adenosine diphosphate (ADP) receptor inhibitors (clopidogrel, prasugrel, ticagrelor, cangrelor) or phosphodiesterase inhibitors (dipyridamole), where the treating physician or patient does not wish to stop these medications,
  7. Concurrent treatment with strong inhibitors of combined CYP3A4 and P-glycoprotein; or strong inducers of CYP3A4,
  8. Any stroke within 1 month prior to enrolment,
  9. Any previous history of a haemorrhagic or lacunar stroke,
  10. Severe heart failure with known ejection fraction <30% or New York Heart Association class III or IV symptoms,
  11. History of hypersensitivity or known contraindication to rivaroxaban,
  12. Uncontrolled hypertension (systolic BP ≥180 mm Hg or diastolic BP ≥110 mm Hg), at the time of screening
  13. Haemoglobin <90 g/L, or platelet count <100 x 109/L,
  14. Significant liver disease (defined as Child-Pugh Class B or C) or Alanine Aminotransferase (ALT) >3 times upper normal limit,
  15. Kidney transplant recipients with a functioning allograft, or scheduled for living-donor kidney transplant surgery,
  16. All countries except Europe: Pregnancy or intention to become pregnant or breast-feeding; Europe only: Women who are not in a postmenopausal state, where postmenopausal is defined as no menses for 12 months without alternative medical causes,
  17. Inability to understand or comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Risk of Major Adverse Cardiac Event (MACE) | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of a composite outcome of;
  * CV death,
  * non-fatal myocardial infarction,
  * stroke, or
  * peripheral artery disease (PAD) events

SECONDARY OUTCOMES:
Composite outcome of cardiovascular death, non-fatal myocardial infarction, or stroke. | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of a composite outcome of cardiovascular death, non-fatal myocardial infarction, or stroke.
Composite outcome of all-cause death, non-fatal myocardial infarction, stroke, or PAD events. | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of a composite of all-cause death, non-fatal myocardial infarction, stroke, or PAD events.
Composite outcome of all-cause death, non-fatal myocardial infarction, or stroke. | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of a composite of all-cause death, non-fatal myocardial infarction, or stroke.
Incidence of Cardiovascular Death | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of Cardiovascular Death
Incidence of Non-Fatal Myocardial Infarction | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of Non-Fatal Myocardial Infarction
Incidence of Stroke | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of Stroke
Incidence of PAD Events | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of PAD events
Net Clinical Benefit - incidence of MACE & Bleeding | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of a composite outcome of cardiovascular death, non-fatal myocardial infarction, stroke, PAD events, fatal bleeding, or symptomatic bleeding into a critical organ.
Incidence of Venous Thromboembolism | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of Venous Thromboembolism

OTHER OUTCOMES:
Cost Effectiveness of Intervention - Cost of intervention, & Net benefit in time to MACE event in intervention, when compared to placebo. | 5 years or trial closure
  To determine whether the intervention, compared to placebo, is cost effective. Where the primary outcome is positive, the cost of providing the intervention will be assessed against the MACE benefit achieved to determine if the treatment meets regulatory guidelines for cost effectiveness. E.g of the Australian Pharmaceutical Benefits Scheme (PBS).
Incidence of Thrombosis of dialysis vascular access | 5 years or trial closure
  To determine whether the intervention, compared to placebo, changes the risk of thrombosis of dialysis vascular access among participants with an arteriovenous fistula/graft.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Badve, Study Chair — The George Institute; Martin Gallagher, Study Chair — The George Institute
Locations (88):
- Australia (11):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Logan Hospital, Meadowbrook, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Bendigo Health, Bendigo, Victoria
  - Sunshine Hospital, St Albans, Victoria
- AZ Sint-Jan Brugge, Bruges, Belgium
- Canada (2):
  - University of Alberta, Edmonton
  - Research St. Joseph's - Hamilton, Hamilton
- France (17):
  - Centre Hospitalier Régional Universitaire de Nancy, Nancy, Meurthe-et-Moselle
  - CH Boulogne-sur-Mer, (CH Boulogne-sur-Mer), Boulogne-sur-Mer
  - Hôpital de la Cavale Blanche, (CHU Brest), Brest
  - AURAL Colmar, (AURAL Colmar), Colmar
  - Hopital Louis Pasteur (CH Colmar), Colmar
  - AURAL Haguenau, (AURAL Haguenau), Haguenau
  - CH Haguenau, (CH Haguenau), Haguenau
  - CH Le Puy-en-Velay, Le Puy-en-Velay
  - Hôpital Edouard Herriot, (CHU Lyon), Lyon
  - Hôpital de la Conception, (AP-HM), Marseille
  - AURAL Mulhouse, (AURAL Mulhouse), Mulhouse
  - CH Mulhouse, (CH Mulhouse), Mulhouse
  - Hôpital Pasteur, (CHU Nice), Nice
  - Hôpital de la Maison Blanche, (CHU Reims), Reims
  - AURAL Strasbourg, (AURAL Strasbourg), Strasbourg
  - Hôpital Bretonneau, (CHRU Tours), Tours
  - Hôpitaux de Brbaois, (ALTIR), Vandœuvre-lès-Nancy
- KRH Klinikum Siloah, Hanover, Germany
- India (21):
  - All India Institute Of Medical Sciences, Raipur, Raipur, Chhattisgarh
  - Muljibhai Patel Urological Hospital, Nadiād, Gujarat
  - Noble Annex Hospital, Hadapsar, Pune Maharashtra
  - All India Institute of Medical Sciences, Bathinda, Bathinda, Punjab
  - Aykai Super Speciality Hospital, Ludhiana, Ludhiana, Punjab
  - Aysha Hospital, Chennai, Tamil Nadu
  - Apollo Hospital, Chennai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Citizens Hospital, Hyderabad, Telangana
  - Nizam's Institute of Medical Sciences, Hyderabad, Hyderabad, Telangana
  - Nutema Hospital, Meerut, Uttar Pradesh
  - AIIMS Bhubaneswar, Bhubaneswar
  - Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh
  - KG Hospital, K.Govindaswamy Naidu Medical Trust, Coimbatore
  - Asian Institute of Nephrology and Urology, Hyderabad
  - VS Hospital, Kilpauk
  - Institute of Post-Graduate Medical Education and Research, Kolkata
  - Nil Ratan Sircar Medical College and Hospital, Kolkata
  - Government Hospital, Nandyāl
  - Safdarjung Hospital, New Delhi
  - Government Hospital, Proddatūr
- Malaysia (11):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz, Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tuanku Ja'afar, Seremban, Seremban, Negeri Sembilan
  - Hospital Raja Permaisuri Bainun, Ipoh, Ipoh, Perak
  - Hospital Seberang Jaya, Seberang Jaya, Pulau Pinang
  - Hospital Queen Elizabeth, Kota Kinabalu, Kota Kinabalu, Sabah
  - Hospital Kajang, Kajang, Selangor
  - Hospital Ampang, Ampang
  - Hospital Pakar Sultanah Fatimah Muar, Muar town
- Tribhuvan University College, Kathmandu, Nepal
- Saudi Arabia (6):
  - Hemodialysis Care Project North Centre, Al Yāsamīn, Riyadh Region
  - Hemodialysis King Abdullah Centre, Al Yāsamīn, Riyadh Region
  - Dialysis Centre - King Abdul Aziz Medical City (KAMC), Ar Rimāyah, Riyadh Region
  - Hemodialysis Care Project South Centre, Riyadh, Riyadh Region
  - King Abdulaziz Medical City - Western Region - Jeddah, Ministry of National Guard - Health Affairs, Jeddah
  - King Saud University Medical City (KSUMC), Riyadh
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
- Taiwan (7):
  - Fu-Jen Catholic University Hospital, Taishan, New Taipei City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City
  - Chung-Shan Medical University Hospital, Taichung
  - Wan fang Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou Medical Center, Taoyuan District
- Tunisia (8):
  - Fattouma Bourguiba Hospital, Monastir
  - Hedi chaker Hospital, Sfax
  - Sahloul Hospital, Sousse
  - Charles Nicolle Hospital, Tunis
  - La Rabta Hospital, Tunis
  - Military Hospital, Tunis
  - Mongi Slim Hospital, Tunis
  - Taher Sfar Hospital, Tunis

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be disseminated in the form of a publication to a relevant clinical journal and presentation at appropriate scientific conferences.
  Individual participant data that underlie the results reported, after de-identification (text, tables, figures, and appendices), may be shared with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: To be confirmed
Access Criteria: * No data should be released that would compromise the trial, unless specifically for safety reasons.
  * There must be a strong scientific or other legitimate rationale for the data to be used for the requested purpose.
  * TRACK Investigators should have a period of exclusivity in which to pursue their aims with the data, before key trial data are made available to other researchers.
  * Adequate resources must be available in order to comply with the request, and the scientific aims of the study must justify the use of such resources.
  * Data release complies with the relevant regulations from all relevant countries.

REFERENCES:
- See also: Trial Website — https://www.tracktrial.org/